CLINICAL TRIAL: NCT03864770
Title: Effectiveness of Extracorporeal Shockwave Therapy on the Patients With Nocturnal Leg Cramps - Possible Related to Myofascial Trigger Point in the Gastrocnemius Muscle
Brief Title: Extracorporeal Shock Wave Therapy Treatment for Nocturnal Leg Cramps
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Li-Wei Chou, Minister of Rehabilitation, China Medical University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMUH108-REC2-006
Record Dates: First submitted 2019-03-05; First posted 2019-03-06 (Actual); Last update posted 2019-03-11 (Actual); Status verified 2019-03

CONDITIONS: Nocturnal Leg Cramps
Keywords: myofascial trigger points; nocturnal leg cramps; extracorporeal shock wave therapy
MeSH Terms: conditions — Sleep-Wake Transition Disorders | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Extracorporeal shock wave therapy and general physical therapy (Experimental): In this arm, the subjects will receive the intervention of extracorporeal shock wave therapy and general physical therapy 3 times a week for 2 weeks, in total 6 times treatments and will be arrange to take efficacy two assessment on 1 week and 2 weeks after 6 times treatments separately.
  Interventions: Device: Extracorporeal shock wave therapy; Procedure: General physical therapy
- Only general physical therapy (Active Comparator): In this arm, the subjects will only receive the intervention of general physical therapy 3 times a week for 2 weeks, in total 6 times treatments and will be arrange to take efficacy two assessment on 1 week and 2 weeks after 6 times treatments separately.
  Interventions: Procedure: General physical therapy

INTERVENTIONS:
Device: Extracorporeal shock wave therapy — Extracorporeal shock wave therapy is a mechanical sound wave that generates energy by extremely high-frequency vibration to compress the medium. Low-energy extracorporeal shock waves can be used for cell regeneration and pain control therapy; medium-high energy can be used to treat patients with poor bone healing; high-energy can be used to lithotrite. In recent years, extracorporeal shock waves have been applied on the musculoskeletal diseases, such as: epicondylitis, plantar fasciitis, chronic pelvic pain, chronic heel pain syndrome, lymphedema, burns, pressure sores, calcific tendinitis and myofascial pain syndrome. This treatment is a non-invasive and safe treatment.
  Arms: Extracorporeal shock wave therapy and general physical therapy
Procedure: General physical therapy — The general physical therapies such as: thermotherapy, straight leg raise (SLR), transcutaneous electrical nerve stimulation (TENS) for treatment on calf muscle.

SUMMARY:
Nocturnal leg cramps (NLCs) are often described as a symptom of sudden and involuntary muscle contraction at night, which often affects sleep quality due to pain and tight discomfort in the thigh, calf and foot. The investigator performed extracorporeal shock wave therapy (ESWT). This experiment used a randomized experiment to assess the immediate, short-term and long-term effects of extracorporeal shock wave therapy on patients with nocturnal leg cramps.

DETAILED DESCRIPTION:
Nocturnal leg cramps (NLCs) are often described as a symptom of sudden and involuntary muscle contraction at night, which often affects sleep quality due to pain and tight discomfort in the thigh, calf and foot. The pathophysiology of nocturnal leg cramps is unclear, but it is generally considered to be associated with excitability lower motor neurons, sleep posture at night, leg muscle fatigue, nerve disability or damage (eg, Parkinson's disease), metabolic diseases (eg : hyperphosphatemia). Generally, quinine or magnesium oxide is the most commonly used pharmacological treatment. The common non-drug treatments are stretching exercise, massage or hot therapy, but there is not enough evidence to indicate which treatment is specific effective.

In a previous study, they proposed that nocturnal leg cramps may be associated with myofascial trigger points (MTrPs) of the gastrocnemius. Other studies have also proposed that extracorporeal shock wave therapy (ESWT) applying to the MTrPs of the upper trapezius muscle could improve cervicogenic headache. We will conduct a randomized parallel study to investigate the efficacy of ESWT on nocturnal leg cramps. Participants will be randomized into two groups: one is only general physical therapy (gPT) and the other one is ESWT + gPT.

The outcome measurement tools including the frequency of nocturnal leg cramps, visual analog scale (VAS), pain pressure threshold (PPT) and muscle tone in the gastrocnemius, range of motion of knee and ankle, and quality of sleep questionnaire were used to compare two groups with regard to the pain intensity, quality of sleep, and overall satisfaction in subjects with nocturnal leg cramps.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 20 y/o patients with NLCs: (1) 4 times/week, last 2 weeks; (2) Occurred in nighttime or resting time of daytime
2. Patients with MTrPs on gastrocnemius (According to the diagnostic criteria proposed by Simons & Travell)

Exclusion Criteria:

1. (1) Taking medication for leg cramps (eg. Quinine, Magnesium oxide); (2) Other drugs that affect research and evaluation (eg. diuretics, statins, calcium channel blockers, anticonvulsants)
2. Congenital lower limb musculoskeletal diseases, Lower limb or spine surgery
3. Uncommunicated or cognitive impaired
4. Patients refused to be recruited

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-03-05 (Estimated); Primary Completion 2019-12-05 (Estimated); Study Completion 2020-02-04 (Estimated)

PRIMARY OUTCOMES:
The frequency of nocturnal leg cramps (FC) | 1 day
  Ask participants to describe the frequency of nocturnal leg cramps (NLCs) in the last week. The frequency of occurrence is recorded on an average of several times a day (times/day). The frequency of nocturnal leg cramps (FC) can be used as a tracking and indicator of treatment.

SECONDARY OUTCOMES:
Visual Analog Scales (VAS) | 1 day
  The visual analogue scale or visual analog scale (VAS) is a psychometric response scale which can be used in questionnaires. This tool used to help a person rate the intensity of certain sensations and feelings, such as pain. A straight line of 100mm is actually marked with 0 mm on the far left and 100mm on the far right. Two faces are drawn on both ends. Explain to the patient that 0 mm means no pain and 100 mm means very painful. From the left end The right shift indicates more and more pain. Take a pen and let the patient draw a short line vertically on the line, representing his painful position, and record the measured cm value. In this test, if the score of the subject decreases, it can represent the treatment is helpful for the improvement of the patient's pain.
Pressure Pain Threshold (PPT) | 1 day
  Pressure pain threshold (PPT) is defined as the minimum force applied which induces pain. This measure has proven to be commonly useful in evaluating tenderness symptom
Range of Motion of knee and ankle joint | 1 day
  Range of motion of knee and ankle joint will be limited when the calf muscle with active myofasical trigger point. To record range of motion of knee and ankle joint for tracking the efficacy of treatment.
Muscle tone | 1 day
  Muscle tone is the muscle's resistance to passive stretch during resting state. The measuring tool called Myotone will calculate three parameters such as tone, elasticity and stiffness automatically and get a value to represent the muscle tone. If the value decrease, it can represent the treatment is helpful for the subjective muscle relax.
Pittsburgh sleep quality index (PSQI) | 1 day
  The Pittsburgh sleep quality index (PSQI) is currently the most effective assessment tool for assessing sleep quality and status in adults. It can be used to assess and track changes in sleep quality after treatment. The Pittsburgh Sleep Quality Assessment (PSQI) content includes (1) subjective sleep quality, (2) sleep latency, (3) sleep duration, (4) sleep efficiency, (5) sleep disturbance, (6) daytime function, and (7) the condition of using sleep pills. The score of the item is from 0 to 3 points, and the total score is from 0 to 21 points. The higher the score means the worse the quality of sleep. If the total score is greater than 5 points that means the poor quality of sleep.

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hawke F, Sadler SG, Katzberg HD, Pourkazemi F, Chuter V, Burns J. Non-drug therapies for the secondary prevention of lower limb muscle cramps. Cochrane Database Syst Rev. 2021 May 17;5(5):CD008496. doi: 10.1002/14651858.CD008496.pub3. PMID 33998664